CLINICAL TRIAL: NCT05440565
Title: Evaluation of Different Colorectal Cancer Screening Strategies: a Prospective Randomized Trial
Brief Title: Evaluation of Different Colorectal Cancer Screening Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2022SDU-QILU-106
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk score (Placebo Comparator)
  Interventions: Diagnostic Test: APCS score
- Fecal immunochemical test (Active Comparator)
  Interventions: Diagnostic Test: Fecal immunochemical test

INTERVENTIONS:
Diagnostic Test: Fecal immunochemical test — Fecal immunochemical test can concentrate the high-risk population.
  Arms: Fecal immunochemical test
Diagnostic Test: APCS score — APCS score can concentrate the high-risk population.
  Arms: Risk score

SUMMARY:
A large-scale randomized controlled trial was conducted to compare different colorectal neoplasms screening strategies.

ELIGIBILITY:
Inclusion Criteria:

* 50-74 years old
* Informed consent is available

Exclusion Criteria:

* Previous colorectal cancer
* Previous colorectal resection
* Previous received cancer-related treatment (except non-melanoma skin cancer)
* Colonoscopy, sigmoidoscopy, CT colonoscopy, and barium enema were performed within 5 years
* Fecal occult blood or fecal DNA was performed within one year
* Symptoms of lower digestive tract diseases requiring colonoscopy include: (1) rectal bleeding occurred more than once in the past 6 months, (2) recorded iron deficiency anemia, and (3) recorded significant weight loss within 6 months (> 10% of baseline weight)
* Suffering from other diseases that affect the benefit of screening or intolerance to colonoscopy (for example, severe pulmonary disease, end-stage renal disease, end-stage liver disease, severe heart failure or recently diagnosed cancer, except non-melanoma skin cancer)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate | up to 30 months
  Detection of intestinal lesions in population